CLINICAL TRIAL: NCT03112447
Title: Treatment of Medial Humeral Epicondyle Fractures in Children With Absorbable Cartilage Nails
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Guoxin Nan, Vice President of Department orthopeadic department, Children's Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHChongqingMU2016
Record Dates: First submitted 2017-03-06; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Fracture Arm
Keywords: medial epicondyle humerus; absorbable cartilage nail

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- absorbable cartilage nail Group (Experimental): 10 males and 7 females, ages 7-15 years (average, 11.8), and 3 patients with elbow dislocation, the fractures were fixed by absorbable cartilage nail
  Interventions: Procedure: absorbable cartilage nail
- traditional Kirschner wire Group (Active Comparator): 10 males and 5 females, ages 8-14 years (average, 12.6), and 4 patients with elbow dislocation, the fractures were fixed by traditional Kirschner wires
  Interventions: Procedure: traditional Kirschner wires

INTERVENTIONS:
Procedure: absorbable cartilage nail — The experiment group patients were fixed with absorbable cartilage nails
  Arms: absorbable cartilage nail Group
Procedure: traditional Kirschner wires — The control group were fixed with traditional Kirschner wires
  Arms: traditional Kirschner wire Group

SUMMARY:
To compare surgical outcomes from medial epicondyle fracture fixation with absorbable cartilage nails to those from traditional Kirschner wire fixation.

DETAILED DESCRIPTION:
From August 2007 to January 2012, 32 patients undergoing surgery for medial humeral epicondyle fractures in our hospital were randomized into group A (traditional Kirschner wire) or group B (absorbable cartilage nail). The same surgical team performed the operations, and patients were followed for over a year. Group A had open reduction with K-wire fixation, and group B was fixed with absorbable cartilage nails. The Bede scoring system was used to evaluate elbow function at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* fractures with more than 2 mm of displacement were treated with cast immobilization

Exclusion Criteria:

* fractures with less than 2 mm of displacement were treated with cast immobilization

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2012-08-01 (Actual); Study Completion 2012-08-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | on 12th month
  Pain Intensity assessed with the Bede Scoring System
Elbow Motion | on 12th month
  Elbow Motion assessed in degrees
Stability | on 12th month
  Stability assessed using the following scoring system: Stable, Moderate Instability, Grossly Unstable.
Elbow Function evaluation | on 12th month
  A specific physician check the patients and ask them to perform the following activity.(comb hair,eat;perform hygiene;don shirt;don shoe)

IPD SHARING:
Plan to Share IPD: No